CLINICAL TRIAL: NCT04258800
Title: Impact of Music During Colonoscopy on Sympathetic - Autonomic Nervous System
Brief Title: Impact of Music in Colonoscopy
Acronym: ColoRelaxTone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: University Hospital Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Professor, Head of Department, University of Ulm
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSIC123
Record Dates: First submitted 2019-12-17; First posted 2020-02-06 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Colonoscopy; Music; Pain
Keywords: colonoscopy; music; relaxation; satisfaction
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With music (Experimental): Colonoscopy performed with music
  Interventions: Device: Music during colonoscopy
- Without music (No Intervention): Colonoscopy performed without music

INTERVENTIONS:
Device: Music during colonoscopy — Music during colonoscopy
  Arms: With music

SUMMARY:
The study examines the impact of music during colonoscopy on sympathetic - autonomic nervous system, whose activity is operationalized by biopotentials signals. The music is chosen by the patients themselves.

The Null hypothesis: The comparison of the sympathetic - autonomic nervous system (operationalized by biopotentials) intensity between colonoscopy "with" vs. "without" music is not significant.

Alternative hypothesis: The comparison of the sympathetic - autonomic nervous system intensity is significantly higher in colonoscopy "without" music vs. "with" music.

DETAILED DESCRIPTION:
In the field of endoscopy, stress and pain play a relevant role before and during the examination. A variety of methods have been evaluated to date to provide the patient with relaxation/distraction during the examination. Especially the use of relaxation music. However, the previous studies refer to a subjective assessment of the participants after the examination. Here at least one potential bias is to be assumed from the post-procedural euphoria through the use of propofol and/or midazolam. Pain reactions express themselves explicitly in autonomous function. In contrast to our previous work, the present study uses biopotential signals for the objective operationalization of stress reduction.

The activity of the sympathetic - autonomic nervous system is operationalized by biopotentials fixed to the body surface:

* in the face area (corrugator, zygomaticus)
* on the hand (skin conductance, temperature)
* on the torso (electrocardiogram) The satisfaction of the patient and endoscopist with endoscopical procedure were asked using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colonoscopy
* conscious sedation with propofol
* ASA state 1 or 2

Exclusion Criteria:

* lack of written informed consent
* pregnancy
* General anaesthetics
* ASA state >2
* deafness, Hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Impact of Music on EMG (M. Zygomaticus, M. Corrugator) | During colonoscopy procedure
  Evaluation of biopotential signals for the objective operationalization of stress reduction
Impact of Music on EKG (heart rate, heart rate variability) | During colonoscopy procedure
  Evaluation of biopotential signals for the objective operationalization of stress reduction
Impact of Music on skin conductance in micro Siemens | During colonoscopy procedure
  Evaluation of biopotential signals for the objective operationalization of stress reduction
Impact of Music on skin temperature in degrees Celsius | During colonoscopy procedure
  Evaluation of biopotential signals for the objective operationalization of stress reduction
Impact of Music on Propofol Dosis in millilitres | During colonoscopy procedure
  Evaluation of sedation requirements for the objective operationalization of stress reduction
Impact of Music on procedure time in minutes | During colonoscopy procedure
  Evaluation of examination time for the objective operationalization of stress reduction
Patient satisfaction with endoscopical procedure by means of questionnaire | Approximately 45 minutes after colonoscopy was finished
  Satisfaction of the patient with endoscopical procedure rated on a scale from 1 to 4 (1 means best rating, 7 means worst rating)
Patient satisfaction with sedation by means of questionnaire | Approximately 45 minutes after colonoscopy was finished
  Satisfaction of the patient with sedation rated on a scale from 1 to 7 (1 means best rating, 7 means worst rating)
Endoscopist satisfaction by means of questionnaire | immediately after colonoscopy was finished
  Satisfaction of the endoscopist with endoscopical procedure rated on a scale from 1 to 7 (1 means best rating, 7 means worst rating)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Walter, MD, Principal Investigator — University Hospital Ulm
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No